CLINICAL TRIAL: NCT03567486
Title: Paraoptic Tumors : Study of the Radiological, Ophthalmological and Intraoperative Predictive Factors of Visual Recovery After Neurosurgical Removal
Brief Title: Predictive Factors of Visual Recovery After Paraoptic Tumors Removal
Acronym: PRONOPTIC
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: DCT_2017_18
Record Dates: First submitted 2018-06-13; First posted 2018-06-25 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Tuberculum Sellae Meningioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Tuberculum sellae meningiomas: Adult patient suffering from tuberculum sellae meningiomas with surgical treatment

SUMMARY:
Paraoptic tumors - including mostly sellar meningiomas, pituitary gland adenomas and craniopharyngiomas - classically affect the visual function. Some preoperative factors, determined on retrospective studies, are known to constitute bad prognostic factors, such as duration of symptoms and retinal nerve fiber layer thinning on OCT. We propose to perform a single center prospective study in which detailed preoperative ophthalmological and radiological criteria will be collected before surgery. Intraoperative information will be noted as well. All these data will be statistically examined regarding the postoperative visual recovery at 3, 6 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* tuberculum sellae meningioma surgical indication

Exclusion Criteria:

* surgical contra indication MRI contra indication optical disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tuberculum sellae meningioma
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
variation of Visual field | between before surgery and 6 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France